CLINICAL TRIAL: NCT05293353
Title: A Prospective Tolerability and Safety Study of a Powdered Human Milk-based Breastmilk Fortifier (Neokare) in Neonates With Gastrointestinal Problems
Brief Title: Neokare Safety and Tolerability Assessment in Neonates With GI Problems
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: University of Southampton (Other); NeoKare Nutrition Ltd (Unknown)
Responsible Party: Sponsor
Other Study IDs: CHI1109
Record Dates: First submitted 2022-02-17; First posted 2022-03-24 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: NEC; Gastroschisis; Intestinal Perforation; Atresia, Intestinal; Hirschsprung Disease; Exomphalos; Volvulus; Anorectal Malformations; Meconium Ileus; Cows Milk Allergy; Preterm
MeSH Terms: conditions — Gastroschisis; Intestinal Perforation; Intestinal Atresia; Hirschsprung Disease; Hernia, Umbilical; Intestinal Volvulus; Anorectal Malformations; Meconium Ileus; Milk Hypersensitivity; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Breast Milk Fortification with NeoKare: Prospective cohort, 50 infants
  Interventions: Other: NeoKare Breast Milk Fortifier
- No Breast Milk Fortification: Retrospective, historical cohort, approx 50 infants

INTERVENTIONS:
Other: NeoKare Breast Milk Fortifier — Powdered product made from human breast milk used to increase nutritional content of mother's own breast milk
  Groups: Breast Milk Fortification with NeoKare

SUMMARY:
With an increasing body of evidence to support a causal link between drinking milk that contain cow's milk protein (CMP) and the development of gastrointestinal disturbance in infants, many clinicians avoid the use of CMP containing feed in high risk babies.

Delivery of adequate nutritional intake is one of the great challenges in the care of newborn infants, particularly those born preterm or with gastrointestinal problems. Whilst there are recognised benefits of human milk, a diet of exclusive human milk may not meet the nutritional demands of the infant. To close this gap, breast milk fortifier (BMF) is typically added to human milk. However, addition of BMF may be associated with gastrointestinal disturbance, possibly due to the fact that it contains CMP.

This research study is to test the tolerability and safety of a new human milk-based BMF in neonates with gastrointestinal problems. It is hoped that this may provide an opportunity for high risk infants, to receive the benefits of human milk whilst minimising the risks reported to be associated with CMP.

Eligible infants will be those in whom nutritional supplementation of breast is deemed clinically necessary, a weight of greater than 1.0kg at the time of starting fortifier and at least one of:

* previous gastrointestinal surgery
* congenital gastrointestinal anomaly
* medically treated gastrointestinal disease
* previously suspected intolerance of CMP based breast milk fortifier in the absence of other gastrointestinal disease

Infants will be started on human milk-based BMF once they are tolerating 100 mls per kilo per day of human breast milk. The human milk-based fortifier will be commenced at half the recommended dose for 48 hours then increase to full strength. This will be continued until the infant reaches 44 weeks corrected gestational age, or until such time as they are deemed to no longer require the additional nutrition.

DETAILED DESCRIPTION:
BACKGROUND There is an increasing body of evidence to support a causal link between ingestion of cow's milk protein (CMP) containing milks and the development of gastrointestinal disturbance in preterm and term infants. In particular the development of necrotising enterocolitis (NEC) has been associated with use of CMP containing feed in both epidemiological studies and a small number of prospective trials. It may be that this is due to a lack of the protective effect of breast milk, rather than CMP pe se. In addition to NEC, CMP containing feed may be implicated in the development of other gastrointestinal disturbance in preterm infants and as such many clinicians avoid the use of CMP containing feed in high risk infants. One such group are preterm infants who have already had an episode of NEC. Others include those born with a congenital anomaly of the gastrointestinal tract such as gastroschisis.

One of the great challenges in the care of the preterm neonate is the delivery of adequate nutritional intake to support growth and development. Whilst there are recognised benefits of human milk for preterm infants, a diet of exclusive human milk does not meet the nutritional and metabolic demands of the preterm infant(4). To close this nutritional gap, breast milk fortifier (BMF) is typically added to human milk. BMF is manufactured from cow's milk, and so contains hydrolysed CMP. However, there is concern that this addition of BMF may be associated with gastrointestinal disturbance, and this may be due to the fact that it contains elements of CMP. In view of this potential association, there is an understandable reluctance to use standard BMF in infants who have already had evidence of gastrointestinal disturbance, such as NEC or gastrointestinal surgery.

RATIONALE Recently a human milk based breast milk fortifier (NeoKare) has become available and is currently being evaluated in the preterm population when compared to current standard feeding practice. Provision of such an exclusive human milk diet may not carry the same risk of gastrointestinal disturbance and may represent an opportunity for high-risk preterm infants that have had NEC, undergone gastrointestinal surgery or had other gastrointestinal disturbance felt to be related to type of milk, to receive the benefits of human milk together with the nutritional benefits of milk fortification, whilst minimising the risks reported to be associated with exposure to CMP. Being able to improve nutrient intakes in this way using human milk based fortifier, may reduce the need for parenteral nutrition, and in turn reduce the risk of complications of parenteral nutrition, length of stay and hospital costs. To date this human milk-based breast milk fortifier has not been formally evaluated in this group of infants.

There is a need to establish if NeoKare is tolerated by infants with pre-existing gastrointestinal disturbance, and see if it can be safely used in this population. There is also a need to see if it enables better nutrition and growth, and earlier cessation of PN, and in turn a shorter length of stay, These may have cost related benefits, which also need to be explored.

Primary objective The primary aim of the study is to investigate the tolerability of a powdered human milk-based breast milk fortifier (Neokare) in infants cared for on a neonatal unit with pre-existing gastrointestinal disturbance (previous gastrointestinal surgery, medically treated gastrointestinal disease, previously suspected intolerance of cow's milk protein-based breast milk fortifier in the absence of other gastrointestinal disease or a congenital gastrointestinal anomaly not requiring surgery). This will be compared to a retrospective control group of similar infants born prior to the study who were not managed using the NeoKare product

Secondary objectives The main secondary aim of the study is to investigate the safety of a powdered human milk-based breast milk fortifier (Neokare) in infants cared for on a neonatal unit with pre-existing gastrointestinal disturbance (previous gastrointestinal surgery, medically treated gastrointestinal disease, previously suspected intolerance of cow's milk protein-based breast milk fortifier in the absence of other gastrointestinal disease or a congenital gastrointestinal anomaly not requiring surgery) This will be compared to a retrospective control group of similar infants born prior to the study who were not managed using the NeoKare product Other secondary aims of the study are to see if, in infants cared for on a neonatal unit with pre-existing gastrointestinal disturbance (previous gastrointestinal surgery, medically treated gastrointestinal disease, previously suspected intolerance of cow's milk protein-based breast milk fortifier in the absence of other gastrointestinal disease or a congenital gastrointestinal anomaly not requiring surgery), the use of a powdered human milk-based breast milk fortifier (Neokare) leads to improvements in growth, nutrition, length of stay, time on parenteral nutrition and other clinical outcomes compared to a retrospective control group of similar infants born prior to the study who were not managed using the NeoKare product. Cost of care will also be compared.

TRIAL DESIGN This will be a Prospective observational cohort study with a retrospective control group

ELIGIBILITY:
Inclusion Criteria:

All of the following must be met:

1. Current weight greater than ≥ 1.5kg (this will reduce to current weight of ≥ 1.0kg following midpoint review if no safety concerns
2. Deemed by attending clinician that fortification of breast milk is desirable either to meet nutritional requirements or optimise growth
3. Exclusive maternal or donor breast milk feeding (at time of starting fortifier)
4. At least one of the following diagnostic criteria:

   1. Any previous gastrointestinal tract surgery. This may include but is not limited:

      * Surgery for NEC
      * Gastroschisis
      * Spontaneous Intestinal Perforation
      * Intestinal Atresias and Webs
      * Malrotation
      * Hirschsprung's disease
      * Volvulus
      * Exomphalos
      * Meconium Ileus/plugs
      * Anorectal anomalies
   2. Medically treated gastrointestinal disease including but not limited to necrotising enterocolitis (based on nationally agreed case definitions), meconium ileus of prematurity (clinical diagnosis), milk curd obstruction (clinical diagnosis)
   3. Previously suspected intolerance of cow's milk protein-based breast milk fortifier in the absence of other gastrointestinal disease (clinical diagnosis)
   4. Congenital gastrointestinal anomaly (not requiring surgery)

Exclusion Criteria:

Any of the following will result in exclusion:

1. Known congenital metabolic disorder
2. Formula fed prior to diagnosis being made
3. Bilateral grade III or IV intra-ventricular haemorrhage
4. Any infant who has had gastrointestinal tract surgery and received feed other than breast milk following surgery and prior to commencing the study
5. Refusal of consent, refusal for the use of pasteurised donor human milk

The reason for these exclusion criteria is to exclude any baby in whom the primary outcome may be adversely influenced by co-existing medical morbidities

Max Age: 44 Weeks | Sex: All
Age Groups: Child
Study Population: The aim of these inclusion criteria is to select a group of babies typically requiring nutritional supplementation of breast milk but in whom there is currently a reluctance to provide cow's milk-based breastmilk fortifiers.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-06-09 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Days of feed intolerance | At 38 weeks postmenstrual age (an average of 8 weeks after initial surgery/gastrointestinal disturbance)
  Defined as number of days enteral feed was withheld for =>12 hours due to concerns about nasogastric aspirate colour or volume, vomiting, abdominal distension, stoma output, stooling or vomiting, as a proportion of the total number of days on which human milk-based breast milk fortifier was included in the feed

SECONDARY OUTCOMES:
Number of adverse events per infant related to the administration of human milk-based breast milk fortifier. | At hospital discharge (an average of 10 weeks after initial surgery/gastrointestinal disturbance)
  Any adverse event felt to be directly related to the administration of human milk-based breast milk fortifier will be determined by the research team and the clinical team caring for the infant.
Mean daily Energy intake between surgery/gastrointestinal disturbance and discharge | At hospital discharge (an average of 10 weeks after initial surgery/gastrointestinal disturbance)
Mean daily protein intake between surgery/gastrointestinal disturbance and discharge | At hospital discharge (an average of 10 weeks after initial surgery/gastrointestinal disturbance)
Mean daily fat intake between surgery/gastrointestinal disturbance and discharge | At hospital discharge (an average of 10 weeks after initial surgery/gastrointestinal disturbance)
Mean daily carbohydrate intake between surgery/gastrointestinal disturbance and discharge | At hospital discharge (an average of 10 weeks after initial surgery/gastrointestinal disturbance)
Mean daily zinc intake between surgery/gastrointestinal disturbance and discharge | At hospital discharge (an average of 10 weeks after initial surgery/gastrointestinal disturbance)
Mean daily selenium intake between surgery/gastrointestinal disturbance and discharge | At hospital discharge (an average of 10 weeks after initial surgery/gastrointestinal disturbance)
Mean daily copper intake between surgery/gastrointestinal disturbance and discharge | At hospital discharge (an average of 10 weeks after initial surgery/gastrointestinal disturbance)
Mean daily vitamin A intake between surgery/gastrointestinal disturbance and discharge | At hospital discharge (an average of 10 weeks after initial surgery/gastrointestinal disturbance)
Mean daily vitamin D intake between surgery/gastrointestinal disturbance and discharge | At hospital discharge (an average of 10 weeks after initial surgery/gastrointestinal disturbance)
Mean daily vitamin E intake between surgery/gastrointestinal disturbance and discharge | At hospital discharge (an average of 10 weeks after initial surgery/gastrointestinal disturbance)
Mean daily vitamin C intake between surgery/gastrointestinal disturbance and discharge | At hospital discharge (an average of 10 weeks after initial surgery/gastrointestinal disturbance)
Mean daily Energy intake whilst on human milk based fortifier | During the intervention period (whilst receiving human milk-based fortifier, an average of 8weeks after initial surgery/gastrointestinal disturbance)
Mean daily protein intake whilst on human milk based fortifier | During the intervention period (whilst receiving human milk-based fortifier, an average of 8weeks after initial surgery/gastrointestinal disturbance)
Mean daily fat intake whilst on human milk based fortifier | During the intervention period (whilst receiving human milk-based fortifier, an average of 8weeks after initial surgery/gastrointestinal disturbance)
Mean daily carbohydrate intake whilst on human milk based fortifier | During the intervention period (whilst receiving human milk-based fortifier, an average of 8weeks after initial surgery/gastrointestinal disturbance)
Mean daily zinc intake whilst on human milk based fortifier | During the intervention period (whilst receiving human milk-based fortifier, an average of 8weeks after initial surgery/gastrointestinal disturbance)
Mean daily selenium intake whilst on human milk based fortifier | During the intervention period (whilst receiving human milk-based fortifier, an average of 8weeks after initial surgery/gastrointestinal disturbance)
Mean daily copper intake whilst on human milk based fortifier | During the intervention period (whilst receiving human milk-based fortifier, an average of 8weeks after initial surgery/gastrointestinal disturbance)
Mean daily vitamin A intake whilst on human milk based fortifier | During the intervention period (whilst receiving human milk-based fortifier, an average of 8weeks after initial surgery/gastrointestinal disturbance)
Mean daily vitamin D intake whilst on human milk based fortifier | During the intervention period (whilst receiving human milk-based fortifier, an average of 8weeks after initial surgery/gastrointestinal disturbance)
Mean daily vitamin E intake whilst on human milk based fortifier | During the intervention period (whilst receiving human milk-based fortifier, an average of 8weeks after initial surgery/gastrointestinal disturbance)
Mean daily vitamin C intake whilst on human milk based fortifier | During the intervention period (whilst receiving human milk-based fortifier, an average of 8weeks after initial surgery/gastrointestinal disturbance)
Growth since study enrollment- weight gain in g/kg/day | At 36 weeks postmenstrual age
Growth since study enrollment- change in weight standard deviation score based on UK reference data | At 36 weeks postmenstrual age
Growth since study enrollment- weight gain in g/kg/day | At Estimated date of delivery
Growth since study enrollment- change in weight standard deviation score based on UK reference data | At Estimated date of delivery
Growth since study enrollment- weight gain in g/kg/day | At hospital discharge (an average of 10 weeks after initial surgery/gastrointestinal disturbance)
Growth since study enrollment- change in weight standard deviation score based on UK reference data | At hospital discharge (an average of 10 weeks after initial surgery/gastrointestinal disturbance)
Growth since study enrollment- weight gain in g/kg/day | At 3 months of age corrected for prematurity
Growth since study enrollment- change in weight standard deviation score based on UK reference data | At 3 months of age corrected for prematurity
Growth since study enrollment- length in mm/week | At 36 weeks postmenstrual age
Growth since study enrollment- change in length standard deviation score based on UK reference data | At 36 weeks postmenstrual age
Growth since study enrollment- length in mm/week | At Estimated date of delivery
Growth since study enrollment- change in length standard deviation score based on UK reference data | At Estimated date of delivery
Growth since study enrollment- length in mm/week | At hospital discharge (an average of 10 weeks after initial surgery/gastrointestinal disturbance)
Growth since study enrollment- change in length standard deviation score based on UK reference data | At hospital discharge (an average of 10 weeks after initial surgery/gastrointestinal disturbance)
Growth since study enrollment- length in mm/week | At 3 months of age corrected for prematurity
Growth since study enrollment- change in length standard deviation score based on UK reference data | At 3 months of age corrected for prematurity
Growth since study enrollment- head circumference in mm/week | At 36 weeks postmenstrual age
Growth since study enrollment- change in head circumference standard deviation score based on UK reference data | At 36 weeks postmenstrual age
Growth since study enrollment- head circumference in mm/week | At Estimated date of delivery
Growth since study enrollment- change in head circumference standard deviation score based on UK reference data | At Estimated date of delivery
Growth since study enrollment- head circumference in mm/week | At hospital discharge (an average of 10 weeks after initial surgery/gastrointestinal disturbance)
Growth since study enrollment- change in head circumference standard deviation score based on UK reference data | At hospital discharge (an average of 10 weeks after initial surgery/gastrointestinal disturbance)
Growth since study enrollment- head circumference in mm/week | At 3 months of age corrected for prematurity
Growth since study enrollment- change in head circumference standard deviation score based on UK reference data | At 3 months of age corrected for prematurity
Number of Episodes of Central Line Associated Blood Stream infection (CLABSI) and NEC during hospital stay after initial initial surgery/gastrointestinal disturbance, defined using existing nationally agreed case definitions | At hospital discharge (an average of 10 weeks after initial surgery/gastrointestinal disturbance)
Days of Parenteral Nutrition (PN) during hospital stay after initial initial surgery/gastrointestinal disturbance, defined as each 24hour period an infants received at least some PN | At hospital discharge (an average of 10 weeks after initial surgery/gastrointestinal disturbance)
Cost of providing PN per day during hospital stay after initial initial surgery/gastrointestinal disturbance | At hospital discharge (an average of 10 weeks after initial surgery/gastrointestinal disturbance)
Number of days spent having level 3 care (according to British Association of Perinatal Medicine criteria with associated tariff cost) during hospital stay after initial initial surgery/gastrointestinal disturbance | At hospital discharge (an average of 10 weeks after initial surgery/gastrointestinal disturbance)
Number of days spent having level 2 care (according to British Association of Perinatal Medicine criteria with associated tariff cost) during hospital stay after initial initial surgery/gastrointestinal disturbance | At hospital discharge (an average of 10 weeks after initial surgery/gastrointestinal disturbance)
Number of days spent having level 1 care (according to British Association of Perinatal Medicine criteria with associated tariff cost) during hospital stay after initial initial surgery/gastrointestinal disturbance | At hospital discharge (an average of 10 weeks after initial surgery/gastrointestinal disturbance)
Number of days spent having 'normal' care (according to British Association of Perinatal Medicine criteria with associated tariff cost) during hospital stay after initial initial surgery/gastrointestinal disturbance | At hospital discharge (an average of 10 weeks after initial surgery/gastrointestinal disturbance)
Number of participants who develop PN associated liver disease stay after initial surgery/GI disturbance-defined as cholestasis (conjugated serum bilirubin 34.2 mmol/L) occurring in the setting of PN, when other specific causes of liver injury excluded | At hospital discharge (an average of 10 weeks after initial surgery/gastrointestinal disturbance)
Length of stay in the hospital (both overall and post-operatively) | At hospital discharge (an average of 10 weeks after initial surgery/gastrointestinal disturbance)
Number of episodes of unplanned gastrointestinal surgery during hospital stay after initial initial surgery/gastrointestinal disturbance | At hospital discharge (an average of 10 weeks after initial surgery/gastrointestinal disturbance)
Number of infants that discontinue fortifier during hospital stay after initial initial surgery/gastrointestinal disturbance | At hospital discharge (an average of 10 weeks after initial surgery/gastrointestinal disturbance)
  The number of infants who have the NeoKare fortifier stopped for clinical reasons. Reason for discontinuation will also be collected
Number of infants who die during the study period and prior to hospital discharge | At hospital discharge (an average of 10 weeks after initial surgery/gastrointestinal disturbance)
Number of episodes of any infections/sepsis requiring antibiotic therapy > 7 days during hospital stay after initial initial surgery/gastrointestinal disturbance | At hospital discharge (an average of 10 weeks after initial surgery/gastrointestinal disturbance)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Johnson, PhD, Principal Investigator — University Hospital Southampton NHS Foundation Trust
Locations (1):
- University Hospital Southampton NHS Foundation Trust, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No